CLINICAL TRIAL: NCT03500861
Title: A Randomized Trial of Trigger Point Dry Needling Versus Sham Needling for Chronic Tension-Type Headache
Brief Title: Trigger Point Dry Needling for Chronic Tension-Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Emine Handan Tüzün, Prof. Dr., Eastern Mediterranean University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ETK00-2017-0121
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Tension-Type Headache; Trigger Points
Keywords: headache characteristics, health-related quality of life.
MeSH Terms: conditions — Tension-Type Headache | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): While the patient was sitting, the therapist firstly cleaned the area with alcohol. Then, DN was applied into the active TrPs on the basis of the technique described by Hong (19). The needle remained in the trigger points for 20 minutes. Upon removal of the needle, the area was compressed firmly with a cotton swab for 60 secs. The DN procedure used sterile stainless-steel acupuncture needles of 0.25x40 mm and 0.25x 25 mm dimensions (Hua Long ®). DN was applied three times a week for 2 weeks, in previously diagnosed active trigger points located in the musculature of the head and the neck.
  Interventions: Other: Dry Needling
- Sham Dry Needling (Sham Comparator): In the Sham Dry Needling (SDN) group, three times a week for 2 weeks, the SDN procedure was applied into the adipose tissue located at any area where an active TrPs was absent.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — The trigger point DN procedure was performed by a certified physiotherapist. While the patient was sitting, the therapist firstly cleaned the area with alcohol. Then, DN was applied into the active TrPs on the basis of the technique described by Hong (19). The needle remained in the trigger points for 20 minutes. Upon removal of the needle, the area was compressed firmly with a cotton swab for 60 secs. The DN procedure used sterile stainless-steel acupuncture needles of 0.25x40 mm and 0.25x 25 mm dimensions (Hua Long ®). DN was applied three times a week for 2 weeks, in previously diagnosed active trigger points located in the musculature of the head and the neck.
  the Sham Dry Needling procedure was applied into the adipose tissue located at any area where an active TrPs was absent.
  Other Names: Sham Dry Needling

SUMMARY:
In this double-blind randomized trial, we aimed to explore the effectiveness of trigger point dry needling in patients with chronic tension type headache (CTTH) in reduction of headache frequency, intensity, duration, and improvement of health-related quality of life (HRQoL).A total of 160 CTTH patients participated in this double-blind, sham-controlled randomized trial. The patients received dry needling using sterile stainless-steel acupuncture needles of 0.25x40 mm and 0.25x 25 mm dimensions three times a week for 2 weeks. The primary outcome measurement which was the headache intensity and, the secondary outcome measurements which were the headache frequency and duration were collected using a headache diary before and after treatment. Another secondary outcome measurement which was the health related quality of life was measured before treatment and at the end of the 1-month follow-up period. HRQoL assessments of patients were performed using Short Form-36 (SF-36). In the dry needling (DN) group, both the primary outcome measurements and the scores of SF-36 subscales were significantly improved after treatment. In the DN group, all effect sizes for headache variables were large. The results of this clinical trial suggest that trigger point dry needling in patients with CTTH is effective and safe in reduction of headache frequency, intensity, duration, and increasing health-related quality of life.

DETAILED DESCRIPTION:
According to the 2013 Global Burden of Disease study, recurrent tension-type headache is the second most common chronic disease worldwide, with an age-standardized prevalence of 21.75 % (1). Although high prevalence of chronic tension-type headache (CTTH) has been reported in all world regions, it is also the most neglected disorder and it leads to headaches that are difficult to treat (2). Myofascial pain can play an important etiologic role. It has been claimed that pain from pericranial head, neck and shoulder muscles is associated with the head and experienced as headache (5, 6). Within the cervical musculature, there are several head and neck muscles, eg. temporal, masseter, upper trapezius, sternocleidomastoid, temporalis, sub-occipital muscles, from which trigger points (TrPs) spread referred pain to the head (6). There are several pharmacological and non-pharmacological therapies for patients with CTTH. Physiotherapy is the most commonly used non-pharmacological treatment of CTTH. Although sports and orthopedic physiotherapists have used dry needling (DN) for a long time to address the pain and dysfunction associated with myofascial trigger points (11), there is insufficient evidence to strongly advocate for use of DN for treatment of CTTH (12). In this double-blind randomized trial, we aimed to explore the effectiveness of trigger point dry needling in patients with CTTH in reduction of headache frequency, intensity, duration, and improve health-related quality of life (HRQoL).

ELIGIBILITY:
Inclusion Criteria:

1. being between 20 and 50 years of age,
2. diagnosed with CTTH according to the International Classification of Headache Disorders-3 (ICHD-3) beta criteria,
3. having at least one active TrP, and
4. having pain intensity greater than 2 cm on the Visual Analog Scale (VAS).

Exclusion Criteria:

1. subjects who have migraine, cluster headache, episodic tension-type headache, secondary headaches and facial pain,
2. subjects who used any medication, except simple analgesics, during treatment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
The headache intensity | Change from baseline headache intensity at the end of 2 weeks and at the end of the 1-month follow-up period.
  On the diary, patients registered the headache intensity, Headache intensity was evaluated using a 10-cm horizontal Visual Analog Scale (cm), (VAS; range: 0 = no pain and 10 = maximum pain)

SECONDARY OUTCOMES:
The headache frequency | Change from baseline headache frequency at the end of 2 weeks and at the end of the 1-month follow-up period.
  On the diary, patients registered the frequency of headaches (days per week)
The headache duration | Change from baseline headache duration at the end of 2 weeks and at the end of the 1-month follow-up period.
  On the diary, patients registered the duration of each headache attack (hours per day).
The quality of life | Change from baseline assessment at the end of the 1-month follow-up period.
  The health related quality of life assessments of patients were performed using the Turkish version of Short Form-36. It includes eight multi-item scales containing between 2 and 10 items each, plus a single item to compare current health with a person's health 1 year ago (health transition). The scales cover the dimensions of physical functioning (PF), role physical (RP), bodily pain (P), general health (GH), vitality (V), social functioning (SF), role emotional (RE), and mental health (MH). All items pertaining to each scale (excluding health transition) are summed and transformed to form a scale from 0 to 100, where a higher score indicates a better state of health or well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Emine H. Tüzün, Prof.Dr., Study Chair — Instructor; Sıla Gildir, MsC., Principal Investigator — Physical Therapist; Goncagül Eroğlu, PT., Principal Investigator — Physical Therapist; Levent Eker, Assist.Prof., Principal Investigator — Instructor
Locations (1):
- 1. Eastern Mediterranean University Health Sciences Faculty, Department of Physiotherapy and Rehabilitation,, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155